CLINICAL TRIAL: NCT07261917
Title: Preoperative Psychotherapy and Its Effects on Anxiety, Hemodynamics, and Pain in Living Kidney Donors
Acronym: PREPSY-KD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Bora Dinc, Associate Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAEK-840
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Living Kidney Donation; Preoperative Anxiety; Postoperative Pain
Keywords: Living kidney donor; Psychiatric intervention; Preoperative anxiety; Postoperative pain; Hemodynamic parameters; Opioid use; Psychological support
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The psychological education and interventions applied to the intervention group were supported by practical and detailed training sessions conducted by a psychiatrist for the anesthesiologist, along with supervision. One hour before the operation, patients underwent a supervised interview lasting approximately 15 minutes under the psychiatrist's supervision upon hospital admission. This interview consisted of history-taking (3-5 minutes), psychoeducation (3-5 minutes), diaphragmatic breathing exercises (1-3 minutes), and guided imagery (3-5 minutes). During the interview, the patient engaged in a conversation, was provided with information about the operation, received standardized psychoeducation about anxiety in collaboration with the psychiatrist, and was guided through anxiety-reducing techniques such as diaphragmatic breathing exercises and guided imagery.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessors (VAS scores) were blinded to the group allocation. Participants, care providers, and investigators were aware of the assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Preoperative Psychiatric Consultation (Experimental): Participants in this group received structured preoperative psychiatric consultation. The intervention consisted of a supervised 15-minute interview conducted one hour before surgery under psychiatrist oversight. The session included history-taking (3-5 minutes), standardized psychoeducation (3-5 minutes), diaphragmatic breathing exercises (1-3 minutes), and guided imagery (3-5 minutes). Psychiatric education and anxiety-reducing techniques were delivered through a standardized protocol supported by training sessions provided to the anesthesiologist.
  Interventions: Behavioral: Preoperative Psychiatric Consultation
- Control Group: Standard Preoperative Care (Active Comparator): Participants in this group received standard preoperative care without psychiatric intervention. Twenty minutes before anesthesia induction, the Beck Anxiety Inventory was administered. Preoperative vital signs, including systolic and diastolic blood pressure, heart rate, and oxygen saturation (SpO2), were recorded in the ward. Intraoperative vital signs were documented before induction, at the 30th minute, and at the 1st hour. During emergence from anesthesia, administered antiemetic and analgesic medications (e.g., paracetamol, tramadol) were documented.
  Interventions: Other: No Intervention: Standard Preoperative Care

INTERVENTIONS:
Behavioral: Preoperative Psychiatric Consultation — A brief psychiatric intervention including psychoeducation, breathing exercises, and guided imagery was provided one hour before surgery under psychiatrist supervision.
  Arms: Intervention Group: Preoperative Psychiatric Consultation
Other: No Intervention: Standard Preoperative Care — Routine preoperative evaluation and intraoperative monitoring without psychiatric intervention.
  Arms: Control Group: Standard Preoperative Care

SUMMARY:
Chronic kidney failure is a condition in which the kidneys progressively lose their ability to filter waste, maintain fluid and electrolyte balance, and support essential physiological functions. When kidney function (glomerular filtration rate, GFR) decreases below 15 ml/min/1.73 m^2, the condition is classified as end-stage renal disease (ESRD), and treatment such as dialysis or kidney transplantation becomes necessary.

Kidney transplantation improves quality of life and survival for individuals with ESRD. However, the transplantation process is physically and psychologically stressful for both recipients and living kidney donors. Preoperative anxiety in donors may adversely affect the surgical process, pain perception, recovery, and overall clinical outcomes.

Psychiatric support prior to surgery may help reduce anxiety and improve physiological stability, pain control, and patient satisfaction during the perioperative period. Such support may also reduce the requirement for analgesic medications and prevent related complications.

This study aims to evaluate the effects of preoperative psychiatric consultation on perioperative anxiety levels, intraoperative hemodynamic parameters, postoperative pain scores, and complication rates in living kidney donors.

DETAILED DESCRIPTION:
Chronic kidney failure is a condition in which the kidneys progressively lose their ability to maintain fluid and electrolyte balance and perform essential endocrine and metabolic functions. This deterioration advances irreversibly due to various underlying diseases. A decrease in GFR below 60 ml/min/1.73 m^2 for more than three months indicates structural and functional abnormalities in the kidneys. When the GFR falls below 15 ml/min/1.73 m^2, the condition is defined as ESRD.

Renal replacement therapy becomes necessary when ESRD develops. Treatment options include lifestyle modifications, medical therapy, hemodialysis, peritoneal dialysis, and kidney transplantation.

Kidney transplantation is an effective treatment modality for patients with ESRD, improving quality of life, supporting long-term survival, and eliminating the need for dialysis. However, this process requires not only physical recovery but also psychological adaptation, involving a prolonged and demanding course.

Kidney transplantation represents a significant source of psychological stress for both donors and recipients. The psychological stress experienced by donors, particularly during the preoperative period, may influence the surgical process and the postoperative recovery period. Elevated preoperative anxiety levels may reduce donor adaptation to the surgical process and adversely affect both psychological and physiological recovery. Psychiatric support, education, and effective anxiety management throughout the surgical process play a critical role in mitigating these negative effects.

High levels of preoperative anxiety may alter pain perception, prolong recovery, and increase the risk of complications. Therefore, reducing preoperative anxiety through psychiatric interventions is essential for helping participants cope with surgical stress and minimizing negative psychological and physiological impacts. Numerous studies have shown that managing anxiety with preoperative psychological support contributes to more stable intraoperative hemodynamic parameters and improved postoperative pain control.

Considering the influence of surgical stress on the inflammatory response in kidney donors, further investigation is required to understand how psychiatric interventions affect these parameters. Psychiatric support also plays an important role in reducing opioid requirements for pain management, minimizing opioid-related side effects, preventing postoperative complications, and enhancing overall patient satisfaction.

This study aims to examine the effects of preoperative anxiety and anxiety-reducing interventions on intraoperative and postoperative hemodynamic parameters, postoperative pain scores, and postoperative complications in living kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* American Society of Anesthesiologists (ASA) physical status Class I-II
* Voluntary participation in the study

Exclusion Criteria:

* Diagnosed diabetes mellitus (DM)
* Development of postoperative delirium
* Previously diagnosed psychiatric disorder or current use of psychiatric medications
* History of analgesic drug use within the last one month
* Diagnosed neurological disorder
* Diagnosed musculoskeletal disorder
* Chronic pain or receiving chronic pain treatment
* Recent severe psychological trauma or relevant psychosocial stressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score | Postoperative 30 minutes, 2 hours, 6 hours, 12 hours, 24 hours, and 48 hours
  Pain severity was measured using a 0-10 Visual Analog Scale (VAS), with 0 indicating no pain and 10 indicating the worst pain imaginable.

SECONDARY OUTCOMES:
State Anxiety Score | 30 minutes before surgery (preoperative), postoperative 24 hours, postoperative 48 hours
  Preoperative and postoperative anxiety levels measured using the Beck Anxiety Inventory (BAI; range 0-63; higher scores indicate greater anxiety).
Postoperative SpO2 Levels | Postoperative 30 minutes, 2 hours, 6 hours, 12 hours, 24 hours, and 48 hours
  Postoperative oxygen saturation (SpO2; %) measured using standard pulse oximetry
Intraoperative Heart Rate | Pre-induction, 30 minutes after induction, and 1 hour after induction
  Intraoperative heart rate measured using standard monitors (beats per minute)
Intraoperative SpO2 Levels | Pre-induction, 30 minutes after induction, and 1 hour after induction
  SpO2 was continuously monitored using standard devices during the intraoperative period at pre-induction, 30 minutes, and 1 hour, and also recorded periodically during the first 48 hours postoperatively.
Intraoperative Systolic Blood Pressure | Pre-induction, 30 minutes after induction, and 1 hour after induction
  Intraoperative systolic blood pressure measured in millimeters of mercury (mmHg)
Intraoperative Diastolic Blood Pressure | Pre-induction, 30 minutes after induction, and 1 hour after induction
  Intraoperative diastolic blood pressure measured in millimeters of mercury (mmHg)
Total Opioid Consumption | Intraoperative period, postoperative first 24 hours
  Total opioid dose administered during and after surgery, recorded in milligrams (mg)
Antiemetic Use | Intraoperative period, postoperative first 6 hours
  Administration of antiemetic agents (e.g., ondansetron), recorded as yes/no and dosage in milligrams (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A final decision regarding sharing of individual participant data (IPD) has not yet been made. IPD sharing will be evaluated after study completion and analysis of the results. If IPD sharing is approved, anonymized datasets will be made available on a publicly accessible repository, and a link will be provided in the "Available IPD/Information" section of the record.

REFERENCES:
- [Background] Sidawy AN, Spergel LM, Besarab A, Allon M, Jennings WC, Padberg FT Jr, Murad MH, Montori VM, O'Hare AM, Calligaro KD, Macsata RA, Lumsden AB, Ascher E; Society for Vascular Surgery. The Society for Vascular Surgery: clinical practice guidelines for the surgical placement and maintenance of arteriovenous hemodialysis access. J Vasc Surg. 2008 Nov;48(5 Suppl):2S-25S. doi: 10.1016/j.jvs.2008.08.042. PMID 19000589
- [Background] Li PK, Chow KM. Peritoneal dialysis patient selection: characteristics for success. Adv Chronic Kidney Dis. 2009 May;16(3):160-8. doi: 10.1053/j.ackd.2009.02.001. PMID 19393965
- [Background] Lv JC, Zhang LX. Prevalence and Disease Burden of Chronic Kidney Disease. Adv Exp Med Biol. 2019;1165:3-15. doi: 10.1007/978-981-13-8871-2_1. PMID 31399958
- [Background] Tola YO, Chow KM, Liang W. Effects of non-pharmacological interventions on preoperative anxiety and postoperative pain in patients undergoing breast cancer surgery: A systematic review. J Clin Nurs. 2021 Dec;30(23-24):3369-3384. doi: 10.1111/jocn.15827. Epub 2021 May 3. PMID 33942405
- [Background] Bayrak A, Sagiroglu G, Copuroglu E. Effects of Preoperative Anxiety on Intraoperative Hemodynamics and Postoperative Pain. J Coll Physicians Surg Pak. 2019 Sep;29(9):868-873. doi: 10.29271/jcpsp.2019.09.868. PMID 31455484
- [Background] Lentine KL, Kasiske BL, Levey AS, Adams PL, Alberu J, Bakr MA, Gallon L, Garvey CA, Guleria S, Li PK, Segev DL, Taler SJ, Tanabe K, Wright L, Zeier MG, Cheung M, Garg AX. KDIGO Clinical Practice Guideline on the Evaluation and Care of Living Kidney Donors. Transplantation. 2017 Aug;101(8S Suppl 1):S1-S109. doi: 10.1097/TP.0000000000001769. PMID 28742762
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT07261917/Prot_SAP_000.pdf